CLINICAL TRIAL: NCT04921059
Title: An Investigation of Heart Rate Recovery Responses to Repeated Active Stand Protocols
Status: Completed | Type: Observational
Sponsor: Caitríona Quinn (Other)
Responsible Party: Sponsor-Investigator, Caitríona Quinn, Research Physiotherapist, St. James's Hospital, Ireland
Organization: St. James's Hospital, Ireland (Other)
Other Study IDs: AS repeatability
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-05

CONDITIONS: Heart Rate Response; Orthostasis
Keywords: Heart rate response; Active Stand
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Active Stand — The participant is asked to lie down for 10 mins without moving or speaking. A heart rate monitor is attached while the participant is lying down. They are then asked to stand up as quickly as possible and to remain standing unassisted for 3 minutes. The participant will be asked to describe any symptoms at 1 and 3 minutes after standing. Blood pressure and heart rate will be monitored constantly throughout the test.

SUMMARY:
Study background:

Impaired heart rate recovery following active stand is associated with morbidity and mortality. Evidence for the repeatability of this measure is limited. This study seeks to determine the repeatability of the active stand procedure in eliciting heart rate recovery in healthy adults of all ages.

Research aims:

The aims of this study are to determine the repeatability of heart rate recovery in response to the active stand procedure among different age groups.

Study design:

This will be a repeatability study with between group comparison.

Study setting:

This study will take place in the Clinical Research Facility in St James's Hospital.

Participants:

Participants will be recruited from the staff and student population of Trinity College Dublin and St James's Hospital, from the Trinity Retirement Association and from the community in the St. James's Hospital catchment area. Participants will be healthy adults (over 18 years old). They will be invited to participate via an email and poster campaign. Participation will be fully voluntary. Participants who meet inclusion criteria will be selected. Informed, explicit voluntary consent will be obtained from each participant.

Data collection and processing:

Data collection and processing will be carried out by the Research Physiotherapist. A clinical visit for the participant will be arranged at a time most convenient for them. Participants will conduct the active stand assessment on three occasions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥18 (considering 18 is the age of legal consent).
* Fluent in English.
* Free of intellectual disability or cognitive impairment that would impair or impede the ability to give informed, explicit consent.
* Free of all exclusion criteria below.

Exclusion Criteria:

* Unstable or un-managed cardiac/respiratory/metabolic conditions (i.e. condition must be diagnosed and being managed as per medical input to be classified as stable and managed).
* Neuro- musculoskeletal disorders.
* Acute musculoskeletal injury or impairment (including acute pain).
* Malignancy.
* Mental illness.
* Chronic infectious disease (Hep C/ HIV/ AIDS).
* Acute systemic infection or illness.
* Taking medication that affects cardiovascular function.
* Exclusion for any other reason deemed appropriate by the research team.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18+ from the staff and students of Trinity College Dublin and St James's Hospital, from the Trinity Retirement Association and from the community in the SJH catchment area.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Baseline Heart Rate | 60 seconds prior to standing assessment
  R-R interval is recorded by portable ECG throughout assessment
Maximum heart rate | Within 3 minutes of standing assessment
  R-R interval is recorded by portable ECG throughout assessment
Minimum heart rate | Within 3 minutes of standing assessment
  R-R interval is recorded by portable ECG throughout assessment

SECONDARY OUTCOMES:
Demographic data | Day 1
  gender, age, relevant past medical history
Height | Day 1
  Centimeters
Weight | Day 1
  Kilograms
Body Mass Index | Day 1
  Kg/m^2
Body Fat Percentage | Day 1
  Percentage
Blood Pressure | At baseline
  Blood Pressure
Vascular Stiffness | Day 1
  Pulse Wave Analysis conducted using the Mobil-O-Graph 24-hour Pulse Wave Analysis (PWA) system.

CONTACTS AND LOCATIONS:
Overall Officials: John Gormley, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Clinical Research Facility, St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared with outside parties.